CLINICAL TRIAL: NCT03903510
Title: A Randomized Control Trial of Virtual Reality to Reduce Anxiety During Pediatric Cast Removal
Brief Title: Virtual Reality During Pediatric Cast Removal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gillette Children's Specialty Healthcare (Other)
Responsible Party: Principal Investigator, Andrew G. Geoergiadis, Pediatric Orthopedic Surgeon, Gillette Children's Specialty Healthcare
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00005315
Record Dates: First submitted 2019-03-27; First posted 2019-04-04 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Fractures, Bone
Keywords: Virtual Reality; Cast removal; Fracture
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Virtual Reality (Experimental): Participants will experience Virtual Reality during their cast removal
  Interventions: Device: Virtual Reality (VR)
- Standard of care (No Intervention): Participants will receive their usual standard of care treatment during cast removal

INTERVENTIONS:
Device: Virtual Reality (VR) — Participants in the experimental group will receive an AppliedVR virtual reality headset during their cast removal.
  Other Names: AppliedVR
  Arms: Virtual Reality

SUMMARY:
This study is a randomized control trial of Virtual Reality during cast removal procedures at a pediatric tertiary care center.

DETAILED DESCRIPTION:
Cast removal is a common outpatient procedure and is a source of pain and anxiety for children. Children are often frightened by the appearance and the noise of the saw. Additionally, the saw blade can become warm, and this can be uncomfortable. Multiple methods have been used and studied to try to make this experience easier for children. These methods include: soft music, therapeutic play, and headphones. Virtual reality (VR) devices are now increasingly affordable and portable. VR could be a way to distract children from the appearance and sound of the procedure. VR has been used in other clinical settings to help patients with the anxiety associated with medical procedures. The investigators propose a randomized trial to assess the responses (e.g. questionnaires and monitors) of children to cast removal with VR versus the standard noise reduction headphones.

ELIGIBILITY:
Inclusion Criteria:

* Sustained a fracture in their arm/leg
* No previous experience with a cast removal
* Must have at least one wrist free of immobilization (for heart rate monitor)
* Parents and patient are English speaking

Exclusion Criteria:

* Patients with a history of epilepsy, ventricular shunt, motion sickness
* Patients with any history of cognitive, visual or hearing impairment

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 184 (Estimated)
Dates: Start 2019-05-21 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline heart rate during cast removal procedure | Heart rate will be measured during the cast removal procedure. As this is a single visit study, heart rate will not be measured at any other time periods throughout the study.
  The change from baseline heart rate during cast removal procedure obtained by using an electronic monitoring wristband and measuring heart rate 15 seconds prior to and continuously during the cast removal procedure.

SECONDARY OUTCOMES:
Change in Parent Reported Wong-Baker FACES Pain Scale Rating | The Wong-Baker FACES Pain Scale assessment will be collected 1 minute prior to and immediately after cast removal.This is a single visit study and the assessment will not be measured at any other time periods.
  Parent reported pain scale that is rated from 0 (minimum) to 10 (maximum), where a higher number indicates increased pain.
Change in Patient Reported Wong-Baker FACES Pain Scale Rating | The Wong-Baker FACES Pain Scale assessment will be collected 1 minute prior to and immediately after cast removal.This is a single visit study and the assessment will not be measured at any other time periods.
  Patient reported pain scale that is rated on a scale of 0 (minimum) to 10 (maximum), where a higher number indicates increased pain.
Visual Analog Scale (VAS): Parental anxiety during cast removal | The VAS anxiety assessment will be performed immediately after the cast removal procedure, which is expected to last 5-10 minutes.This is a single visit study and the assessment will not be measured at any other time periods.
  Parental anxiety will be self reported using a 0 (minimum) to 100 (maximum) scale, where a higher number indicates increased anxiety.
Visual Analog Scale (VAS): Patient anxiety during cast removal | The VAS anxiety assessment will be performed immediately after the cast removal procedure, which is expected to last 5-10 minutes.This is a single visit study and the assessment will not be measured at any other time periods.
  Patient anxiety regarding the cast removal will be self reported using a 0 (minimum) to 100 (maximum) scale, where a higher number indicates increased anxiety.
Visual Analog Scale (VAS): Parental Satisfaction | The VAS parental satisfaction assessment will be performed immediately after the cast removal procedure, which is expected to last 5-10 minutes.This is a single visit study and the assessment will not be measured at any other time periods.
  Parental satisfaction regarding the cast removal will be self reported using a 0 (minimum) to 100 (maximum) scale, where a higher number indicates increased satisfaction.
Visual Analog Scale (VAS): Parental Assessment of Pleasantness | The VAS parental satisfaction assessment will be performed immediately after the cast removal procedure, which is expected to last 5-10 minutes.This is a single visit study and the assessment will not be measured at any other time periods.
  Parental report of how pleasant the cast removal was. Self reported using a 0 (minimum) to 100 (maximum) scale, where a higher number indicates increased pleasantness.
Visual Analog Scale (VAS): Parent Reported Worst Pain During Treatment | The VAS parental worst pain assessment will be performed immediately after the cast removal procedure, which is expected to last 5-10 minutes.This is a single visit study and the assessment will not be measured at any other time periods.
  Parental report of the highest level of pain experienced by the child during the cast removal. Reported using a 0 (minimum) to 100 (maximum) scale, where a higher number indicates increased pain.
Visual Analog Scale (VAS): Patient Reported Worst Pain During Treatment | The VAS patient worst pain assessment will be performed immediately after the cast removal procedure, which is expected to last 5-10 minutes.This is a single visit study and the assessment will not be measured at any other time periods.
  Patient report of the highest level of pain experienced by the child during the cast removal. Reported using a 0 (minimum) to 100 (maximum) scale, where a higher number indicates increased pain.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G Georgiadis, MD, Principal Investigator — Pediatric Orthopedic Surgeon
Locations (1):
- Gillette Children's Specialty Healthcare, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naranje SM, Erali RA, Warner WC Jr, Sawyer JR, Kelly DM. Epidemiology of Pediatric Fractures Presenting to Emergency Departments in the United States. J Pediatr Orthop. 2016 Jun;36(4):e45-8. doi: 10.1097/BPO.0000000000000595. PMID 26177059
- [Background] Wiggins CE, Brown KD. Hearing protection and cast saw noise. J South Orthop Assoc. 1996 Spring;5(1):1-4. PMID 8673584
- [Background] Katz K, Fogelman R, Attias J, Baron E, Soudry M. Anxiety reaction in children during removal of their plaster cast with a saw. J Bone Joint Surg Br. 2001 Apr;83(3):388-90. doi: 10.1302/0301-620x.83b3.10487. PMID 11341425
- [Background] Post JM, Switzer KD, Brown DK, Meinzen-Derr J, Dively J, Dunkin BS, Mehlman CT. Cast saw noise does not reach occupational hazard levels. J Pediatr Orthop. 2013 Jul-Aug;33(5):580-4. doi: 10.1097/BPO.0b013e318288b5e4. PMID 23752160
- [Background] Liu RW, Mehta P, Fortuna S, Armstrong DG, Cooperman DR, Thompson GH, Gilmore A. A randomized prospective study of music therapy for reducing anxiety during cast room procedures. J Pediatr Orthop. 2007 Oct-Nov;27(7):831-3. doi: 10.1097/BPO.0b013e3181558a4e. PMID 17878794
- [Background] Wong CL, Ip WY, Kwok BMC, Choi KC, Ng BKW, Chan CWH. Effects of therapeutic play on children undergoing cast-removal procedures: a randomised controlled trial. BMJ Open. 2018 Jul 5;8(7):e021071. doi: 10.1136/bmjopen-2017-021071. PMID 29980545
- [Background] Carmichael KD, Westmoreland J. Effectiveness of ear protection in reducing anxiety during cast removal in children. Am J Orthop (Belle Mead NJ). 2005 Jan;34(1):43-6. PMID 15707139
- [Background] Mahan ST, Harris MS, Lierhaus AM, Miller PE, DiFazio RL. Noise Reduction to Reduce Patient Anxiety During Cast Removal: Can We Decrease Patient Anxiety With Cast Removal by Wearing Noise Reduction Headphones During Cast Saw Use? Orthop Nurs. 2017 Jul/Aug;36(4):271-278. doi: 10.1097/NOR.0000000000000365. PMID 28737634
- [Background] Hoffmann C. COX-2 in brain and spinal cord implications for therapeutic use. Curr Med Chem. 2000 Nov;7(11):1113-20. doi: 10.2174/0929867003374282. PMID 11032961
- [Background] Gold JI, Kim SH, Kant AJ, Joseph MH, Rizzo AS. Effectiveness of virtual reality for pediatric pain distraction during i.v. placement. Cyberpsychol Behav. 2006 Apr;9(2):207-12. doi: 10.1089/cpb.2006.9.207. PMID 16640481
- [Background] Asl Aminabadi N, Erfanparast L, Sohrabi A, Ghertasi Oskouei S, Naghili A. The Impact of Virtual Reality Distraction on Pain and Anxiety during Dental Treatment in 4-6 Year-Old Children: a Randomized Controlled Clinical Trial. J Dent Res Dent Clin Dent Prospects. 2012 Fall;6(4):117-24. doi: 10.5681/joddd.2012.025. Epub 2012 Nov 12. PMID 23277857
- [Background] Nilsson S, Finnstrom B, Kokinsky E. The FLACC behavioral scale for procedural pain assessment in children aged 5-16 years. Paediatr Anaesth. 2008 Aug;18(8):767-74. doi: 10.1111/j.1460-9592.2008.02655.x. PMID 18613934
- [Background] Steele E, Grimmer K, Thomas B, Mulley B, Fulton I, Hoffman H. Virtual reality as a pediatric pain modulation technique: a case study. Cyberpsychol Behav. 2003 Dec;6(6):633-8. doi: 10.1089/109493103322725405. PMID 14756928
- [Background] Hoffman HG, Doctor JN, Patterson DR, Carrougher GJ, Furness TA 3rd. Virtual reality as an adjunctive pain control during burn wound care in adolescent patients. Pain. 2000 Mar;85(1-2):305-9. doi: 10.1016/s0304-3959(99)00275-4. PMID 10692634
- [Background] Hoffman HG, Patterson DR, Carrougher GJ. Use of virtual reality for adjunctive treatment of adult burn pain during physical therapy: a controlled study. Clin J Pain. 2000 Sep;16(3):244-50. doi: 10.1097/00002508-200009000-00010. PMID 11014398
- [Background] Sharar SR, Miller W, Teeley A, Soltani M, Hoffman HG, Jensen MP, Patterson DR. Applications of virtual reality for pain management in burn-injured patients. Expert Rev Neurother. 2008 Nov;8(11):1667-74. doi: 10.1586/14737175.8.11.1667. PMID 18986237
- [Background] Hoffman HG, Seibel EJ, Richards TL, Furness TA, Patterson DR, Sharar SR. Virtual reality helmet display quality influences the magnitude of virtual reality analgesia. J Pain. 2006 Nov;7(11):843-50. doi: 10.1016/j.jpain.2006.04.006. PMID 17074626
- [Background] Schmitt YS, Hoffman HG, Blough DK, Patterson DR, Jensen MP, Soltani M, Carrougher GJ, Nakamura D, Sharar SR. A randomized, controlled trial of immersive virtual reality analgesia, during physical therapy for pediatric burns. Burns. 2011 Feb;37(1):61-8. doi: 10.1016/j.burns.2010.07.007. Epub 2010 Aug 7. PMID 20692769
- [Background] Hoffman HG, Sharar SR, Coda B, Everett JJ, Ciol M, Richards T, Patterson DR. Manipulating presence influences the magnitude of virtual reality analgesia. Pain. 2004 Sep;111(1-2):162-8. doi: 10.1016/j.pain.2004.06.013. PMID 15327820